CLINICAL TRIAL: NCT01486394
Title: Focused Sonographic Examination of the Heart, Lungs and Deep Veins in an Unselected Population of Acute Admitted Patients With Respiratory Symptoms: a Randomised Clinical Trial
Brief Title: Sonography in an Unselected Population of Acute Admitted Patients With Respiratory Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Borbjerg Laursen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S-2010074
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Dyspnoea; Chest Pain; Cough
MeSH Terms: conditions — Dyspnea; Chest Pain; Cough

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Focused sonography (Experimental): Intervention group: After the primary evaluation by a physician in the emergency department, focused sonography of the patients heart, lungs and deep veins in the legs are performed. Hereafter the further examinations and treatment are done according to hospital guidelines.
  Interventions: Other: Focused Sonography of the heart, lungs and deep veins
- Usual treatment and diagnostic work-up (No Intervention): Control group: After the primary evaluation by a physician in the emergency department. Hereafter the further examinations and treatment are done according to hospital guidelines.

INTERVENTIONS:
Other: Focused Sonography of the heart, lungs and deep veins — The patient is randomised to either a control group where usual treatment and diagnostic work-up is performed or to an intervention group where usual treatment and diagnostic workup are supplemented by a sonographic examination of the heart, lungs and deep veins are performed within one hour after the primary evaluation. The primary evaluation is defined as the first evaluation of the patient by a physician in the Acute Medical Admission Department.
  Arms: Focused sonography

SUMMARY:
The purpose of this study is to determine whether focused sonography of the heart, lungs and deep veins can increase the number of patients with respiratory symptoms correctly diagnosed in an emergency department.

ELIGIBILITY:
Inclusion criteria:

All 4 of the following must be present:

1. The sonographic examination can be performed before or within 1 hour after the primary evaluation
2. Patient is 18 years or older
3. Patient able and willing to give informed consent
4. One ore more of the following symptoms or clinical findings at admission to the emergency department

   * Respiratory rate > 20 breaths per minute
   * Saturation < 95%
   * Oxygen therapy initiated
   * The patient has a principal complaint of dyspnoea
   * The patient has a principal complaint of coughing
   * The patient has a principal complaint of chest pain

Exclusion Criteria:

One of the following:

1. The sonographic examination can not be performed within 1 hour after the primary evaluation
2. The patient is 17 years or younger
3. The patient not able or willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The number of patients with a correct presumptive diagnosis within 4 hours after hospital admission. | 4 hours after hospital admission
  The 4-hour presumptive diagnosis are compared to the final diagnosis obtained by audit after the patient has been discharged from the hospital (gold standard).

SECONDARY OUTCOMES:
Number of patients with a correct presumptive diagnosis after primary evaluation in the control group and after sonography in the intervention group. | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Sensitivity, specificity, positive predictive values, negative predictive values and diagnostic accuracy of the primary evaluation and the "4-hour" presumptive diagnosis. | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Number of patients receiving appropriate, inappropriate and no specific treatment 4-hours after admission | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
30 day mortality | 30 days after the patient has been admitted to the hospital
In-hospital mortality | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Number of patients transferred to an intensive care unit | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Number of patients given an appropriate, inappropriate and no specific treatment after primary evaluation in the control group and after sonography in the intervention group | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Time to diagnostic / therapeutic thoracocentesis | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks
Length of hospital stay | Participants will be followed for the duration of the hospital stay, an expected range of up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Laursen, M.D, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Laursen CB, Sloth E, Lassen AT, Christensen Rd, Lambrechtsen J, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Point-of-care ultrasonography in patients admitted with respiratory symptoms: a single-blind, randomised controlled trial. Lancet Respir Med. 2014 Aug;2(8):638-46. doi: 10.1016/S2213-2600(14)70135-3. Epub 2014 Jul 3. PMID 24998674
- [Derived] Laursen CB, Sloth E, Lassen AT, Christensen RD, Lambrechtsen J, Madsen PH, Henriksen DP, Davidsen JR, Rasmussen F. Focused sonographic examination of the heart, lungs and deep veins in an unselected population of acute admitted patients with respiratory symptoms: a protocol for a prospective, blinded, randomised controlled trial. BMJ Open. 2012 May 30;2(3):e001369. doi: 10.1136/bmjopen-2012-001369. Print 2012. PMID 22649177